CLINICAL TRIAL: NCT06642844
Title: Bevacizumab-based Chemotherapy Tailored to the Pharmacokinetics of Bevacizumab in First-line Treatment of Unresectable Metastatic Colorectal Cancer: a Randomized, Multicenter, Double-blind Phase 3 Study
Brief Title: Bevacizumab-based Chemotherapy Adapted to Bevacizumab Pharmacokinetics in 1st-line Treatment
Acronym: PHARBEVACOL
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: CHU DE BESANCON (Unknown); Gustave Roussy, Cancer Campus, Grand Paris (Other); CHU de Clermont-Ferrand (Unknown); CHU de Reims (Other); CHU de Brest (Unknown); AP-HP, Hôpital Pitié- Salpétrière (Unknown); University Hospital, Rouen (Other); Poitiers University Hospital (Other); Institut Paoli-Calmettes (Other); Rennes University Hospital (Other); University Hospital, Toulouse (Other); AP-HP, Hôpital Saint-Louis (Unknown); HCL Hôpital Edouard Hériot (Unknown); Centre Hospitalier Universitaire Dijon (Other); Nantes University Hospital (Other); Centre Hospitalier Universitaire, Amiens (Other); Hôpital Privé Jean Mermoz (Unknown); AP-HP, Hôpital Henri Mondor (Unknown); AP-HP, Hôpital Paul Brousse (Unknown); CHG de St-Malo (Unknown); Polyclinique de Blois (Unknown); University Hospital, Caen (Other); Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR230009
Record Dates: First submitted 2024-03-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Unresectable Metastatic Colorectal Cancer
MeSH Terms: interventions — Bevacizumab; Control Groups

STUDY DESIGN:
Intervention Model Description: This project is a multicenter, double-blind, randomized trial in two parallel groups.
Who Masked: Participant, Investigator
Masking Description: Double blinding (patients and investigators) will be applied to this trial with respect to the dose of bevacizumab administered throughout the study, except in specific circumstances such as in emergency cases, and only if knowledge of the dose is likely to influence management.
  The dose of bevacizumab will be administered in 2 preparations and in the following order:
  * 1. Preparation at 5 mg/kg, open label;
  * 2. Preparation at 5 mg/kg or placebo, blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Group A (Experimental): Patients randomized to the experimental group of the trial will receive bevacizumab as an IV infusion at a dose of 10 mg/kg, administered in 2 preparations of 5 mg/kg, every 2 weeks. Patients will receive treatment until progression, patient refusal, or unacceptable toxicity.
  Interventions: Drug: Avastin, 25 Mg/mL Intravenous Solution
- Active comparator: Group B (Active Comparator): Patients randomized to the control group of the trial will receive bevacizumab at a dose of 5 mg/kg and placebo (NaCl) every two weeks. Patients will receive treatment until progression, patient refusal, or unacceptable toxicity.
  Interventions: Drug: Avastin, 25 Mg/mL Intravenous Solution

INTERVENTIONS:
Drug: Avastin, 25 Mg/mL Intravenous Solution — Experimental group/ Patients randomized to the experimental group of the trial will receive bevacizumab as an IV infusion at a dose of 10 mg/kg, administered in 2 preparations of 5 mg/kg, every 2 weeks. Patients will receive treatment until progression, patient refusal, or unacceptable toxicity.
  Control group: Patients randomized to the control group of the trial will receive bevacizumab at a dose of 5 mg/kg and placebo (NaCl) every two weeks. Patients will receive treatment until progression, patient refusal, or unacceptable toxicity.
  Other Names: Experimental group; Control group

SUMMARY:
Bevacizumab is a standard drug for metastatic colorectal cancer (mCRC) in combination with cytotoxic chemotherapy. However, inter-individual pharmacokinetic variability was observed for bevacizumab and an exposure-response relationship for efficacy was described for bevacizumab in mCRC patients treated with 1st-line bevacizumab-based chemotherapy.

DETAILED DESCRIPTION:
The primary objective is to evaluate the effect of doubling the dose of bevacizumab in mCRC patients whose initial serum bevacizumab concentration is ≤15.5 mg/L on progression-free survival (PFS).

This project is a multicenter, double-blind, randomized trial in two parallel groups.

The primary endpoint is progression-free survival (PFS)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years.
* Histologically proven metastatic colorectal adenocarcinoma (on primary tumor and/or metastases) inoperable, well documented, i.e. not compatible with complete oncological resection at inclusion.
* For whom treatment with bevacizumab is indicated.
* For women of childbearing age: effective contraception.
* ECOG Performance status (PS) 0-2.
* No prior treatment of metastatic disease (in the case of adjuvant treatment, interval between the end of chemotherapy and relapse > 6 months if fluoropyrimidine alone or > 12 months if FOLFOX).
* At least one evaluable or measurable lesion assessed by computed tomography (CT) according to RECIST v1.1 criteria.
* Life expectancy greater than 3 months.
* Adequate hematological, renal and hepatic biological parameters: neutrophils ≥ 1.5x109/L; platelets ≥ 100x109/L; hemoglobin ≥ 9 g/dL; serum creatinine <150 μmol/L; bilirubinemia ≤ 1.5 x upper limit of normal (ULN), alkaline phosphatase < 5xULN; proteinuria < 2+ (urine dipstick) or ≤ 1 g/24h.
* Written informed consent signed by the patient.
* Patient affiliated to a French social security system.

Randomization criteria in the experimental phase:

- Serum concentration of bevacizumab on D14 ≤ 15.5 mg/L (measured just before the 2nd infusion of bevacizumab).

Exclusion Criteria:

Less than 6 months from the end of any prior chemotherapy, radiotherapy or adjuvant surgery.

* Patient with a known non-indication or contraindication to first-line chemotherapy based on bevacizumab.
* Cardiovascular contraindication to the prescription of bevacizumab: heart failure, cardiovascular event within 6 months, NYHA ≥ 2 (New York Heart Association), poorly controlled arterial hypertension, history of hypertensive crisis or hypertensive encephalopathy; Grade 3/4 anterior venous thromboembolism (NCI-CTCAE)
* Inadequate hematological, hepatic and renal function
* Urine test strip for proteinuria ≥ 2+ unless proteinuria < 1 g / 24 hours is demonstrated.
* Current or recent (within 10 days of study enrollment) use of aspirin (>325 mg/day) or clopidogrel (>75 mg/day).
* Current or recent use (within 10 days before the first dose of bevacizumab) of oral or parenteral therapeutic anticoagulants or thrombolytic agents for therapeutic purposes.
* Untreated CNS metastases or treatment of brain metastases, either by surgical or radiological techniques, must have been completed more than 4 weeks before the first study treatment.
* Surgical procedure (including open biopsy, surgical resection, wound revision, or other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to study enrollment or anticipation of study need for major surgery during the study.
* Serious non-healing wound, active ulcer or untreated bone fracture.
* Other neoplasias (previous or current), except:

  * i/ carcinoma in situ of the cervix adequately treated,
  * ii/ basal cell or squamous cell carcinoma of the skin,
  * iii/ cancer in complete remission for more than 5 years.
* Other illnesses, which, according to the doctor, are life-threatening to the patient and/or which are uncontrolled.
* Primary tumor in place and symptomatic (occlusion, hemorrhage).
* Pregnant or breastfeeding women.
* Patients unable to give consent.
* Patients under guardianship, curatorship or legal protection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is progression-free survival (PFS) | up to death
  The SS was defined as the time interval for randomized patients between the date of start of treatment and date of first clinical and/or radiological progression or death whatever the cause, in depending on what survives first.of first clinical and/or radiological progression or death whatever the cause, in depending on what survives first.progression (PD) per RECIST 1.1 or death due to any cause, whichever occurs first. A patient alive without progression will be censored on the date from the last follow-up visit.

SECONDARY OUTCOMES:
Safety profile | Up to approximately 10 months
  Number of Participants Who Experienced an Adverse Event (AE) per NCI-CATCAE5.0 classification
Overall Survival (OS) | Up to approximately 25 months
  OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of analysis were censored at the date of last known contact.
Best Overall Response Rate (BORR) Per RECIST1.1 | Up to approximately 10 months
  BORR is defined as the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started) assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions). Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Depth of response (DpR) | Up to approximately 10 months
  DpR was defined as the relative change in the sum of the target lesions' longest diameters at their smallest attained sizes compared to baseline time.
rate of secondary resection of metastases | Up to approximately 10 months
  secondary resection of initially unresectable metastases of colorectal cancer
Patient quality of life | Up to approximately 10 months
  Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 and European Quality of Life 5 Dimensions 5 Level Version questionnaires
  Measure Description:
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 30 questions are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores meant a better level of function.
  The EQ-5D-5L is a generic tool for Patient-Reported Outcomes (PRO) measurement using 6 5 questions that can assess patients' quality of life, irrespective of the disease. .
  It includes a vertical EQ visual analog scale (EQ VAS, 0-100 points)
Serum concentrations of bevacizumab | on day 14 of the first administration, and at 2 months from randomization (= 3 months from the first course)
  Serum concentrations of bevacizumab in order to evaluate the effect of doubling the administered dose of bevacizumab.
Medical-economic analysis | up to death
  A model-based cost-effectiveness analysis will be performed for estimating the Incremental Cost-Utility Ratio (cost per QALY gained) et the Incremental Cost-Effectiveness Ratio (cost per life-year gained) from the Healthcare system perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Borg, Principal Investigator — Besançon, FRANCE; Michel Ducreux, Principal Investigator — Gustave Roussy, FRANCE; Caroline Petorin, Principal Investigator — Clermont-Ferrand, FRANCE; Olivier Bouché, Principal Investigator — Reims, FRANCE; Jean-Philippe Metges, Principal Investigator — Brest, FRANCE; Jean-Baptiste Bachet, Principal Investigator — Pitié- Salpétrière, FRANCE; Frédéric Di Fiore, Principal Investigator — Rouen, FRANCE; David Tougeron, Principal Investigator — Poitiers, FRANCE; Astrid Lièvre, Principal Investigator — Rennes, FRANCE; Rosine Guimbaud, Principal Investigator — Toulouse , FRANCE; Thomas Aparicio, Principal Investigator — St Louis , FRANCE; Thomas Walter, Principal Investigator — Edouard Hériot, FRANCE; Côme Lepage, Principal Investigator — Dijon, FRANCE; Yann Touchefeu, Principal Investigator — Nantes, FRANCE; Vincent Hautefeuille, Principal Investigator — Amiens, FRANCE; Pascal Artru, Principal Investigator — Jean Mermoz, FRANCE; Christophe Tournigand, Principal Investigator — Henri Mondor, France; Pascal Hammel, Principal Investigator — Paul Brousse, FRANCE; Romain Desgrippes, Principal Investigator — St-Malo, FRANCE; Philippe Laplaige, Principal Investigator — Blois, FRANCE; Karine Bouhier-Leporrier, Principal Investigator — Caen, FRANCE; Marie Muller, Principal Investigator — Nancy, france